CLINICAL TRIAL: NCT04468243
Title: A Nurse-led Intervention in Patients With Newly Diagnosed Cancer and Type 2 Diabetes: A Pilot RCT Feasibility Study
Brief Title: Pilot RCT Feasibility Study: Cancer and T2D
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201902145; OCR35482 (Other: University of Florida)
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 2; Cancer
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led (Experimental): Nurse-led (group A). Patients randomized to group A will be taken to an available consultation room within the clinic and provided brief diabetes education which includes understanding what it means to have diabetes, healthy eating, and physical activity. Patients will also receive instructions on how to use a glucometer and how to take Metformin.
  Interventions: Other: Nurse-led diabetes care
- Usual Care (No Intervention): Usual Care (Control; group B). Patients randomized to usual care will be informed of their HbA1c value, will continue to receive usual cancer care, and will be encouraged to follow-up with their PCP for T2D management. The RA will ensure that oncology visit clinic notes and the results of the HbA1c testing are relayed to the patient's PCP office. Patients who do not have a PCP identified will be referred to an appropriate provider.

INTERVENTIONS:
Other: Nurse-led diabetes care — Nurse-led brief diabetes education, instructions on glucometer and Metformin use, patients receive prescriptions for Metformin and blood glucose testing kit
  Arms: Nurse-led

SUMMARY:
The purpose of this study is to test a nurse-led intervention for adults with newly diagnosed cancer and undiagnosed/newly diagnosed Type-2 diabetes

DETAILED DESCRIPTION:
Specific Aim 1: To examine study feasibility of a nurse-led intervention for adults with newly diagnosed cancer and T2D. We define feasibility indicators as: (a) efficient study recruitment is possible given prevalence of T2D (diagnosed and undiagnosed) in UF patients with newly diagnosed cancer; (b) retention rates in both groups ≥80% to indicate that the study design and methods are adequately patient-centered; (c) identified barriers to and facilitators of a nurse-led intervention are respectively modifiable or optimizable; and (d) patient acceptability scores >8 for the study procedures. We hypothesize that we will recruit up to 40 patients within 18 months and retain ≥ 80% of patients in all groups; minor but important revisions will be required to resolve issues identified with using the nurse-led intervention; and 80% of patients from both groups who complete the study will report that the burden of the study is acceptable through their retention in the study.

Specific Aim 2: To determine the variation in HbA1c at baseline and at the end of the three-month intervention period in each of the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* a) 18 years and older
* b) Using pathology reports, a new diagnosis of a solid tumor cancer or lymphoma within the past 3 months
* c) Patients being treated with curative intent or those with a prognosis estimated to be >2 years, as best assessed by the oncologist.
* d) First medical oncology outpatient visit at UF within the past 3 months
* e) Plans to continue cancer care at UF
* f) Speaks and reads English
* g) Can comply with study related procedures, per the treating oncologist or advanced practice provider

Exclusion Criteria:

* a) Diagnosis of leukemia or pancreatic cancer as the new cancer diagnosis
* b) Being treated for T2D for > than 3 months
* c) eGFR <45mL/minute/1.73m2
* d) Liver insufficiency (defined as liver enzymes over 5 times the upper limit of normal or clinical sequelae of advanced cirrhosis as documented by the treating oncologist or Advanced Practice Providers.
* e) Active infection requiring systemic antibiotics
* f) Taking systemic steroids of more than 1-week duration. Must have stopped >3 days prior to study enrollment. Note, inhaled or topical steroids are not exclusion criteria.
* g) Planning to receive cancer care at a location outside of UF
* h) Enrolled in another study with similar outcomes.
* i) Currently taking metformin or known inability to tolerate it

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Acceptability | At 3-month study visit
  Study acceptability (scores>8 indicate adequate acceptability) will be measured via the Study Acceptability Scale questionnaire for both groups
Point of Care HbA1c Test | At baseline visit and at 3-month study visit
  To determine the variation in HbA1c at baseline and at the end of the three-month intervention period in each of the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Scarton, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No